CLINICAL TRIAL: NCT00397319
Title: The Role of Growth Hormone in Cardiovascular Health
Brief Title: Growth Hormone's Effect on the Cardiovascular System
Status: Terminated | Type: Observational
Why Stopped: Inadequate retention of GHD adults to maintain power to study the effect of GH on fibrinolysis. A comparison between GHD adults and controls was completed.
Sponsor: Vanderbilt University (Other)
Collaborators: Pfizer (Industry); National Center for Research Resources (NCRR) (NIH)
Other Study IDs: 050045; 1422
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2007-07-03 (Estimated); Status verified 2007-07

CONDITIONS: Growth Hormone Deficiency
Keywords: Growth Hormone; Cardiovascular System
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Growth Hormone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Drug: Growth Hormone

SUMMARY:
To evaluate specific markers of cardiovascular risk before and after growth hormone replacement therapy in a population of growth hormone deficient adults, as compared to an age, gender, and BMI-matched healthy population.

DETAILED DESCRIPTION:
Growth hormone deficiency (GHD) is associated with increased cardiovascular morbidity and mortality. The effects of such a deficiency include decreased exercise capacity and tolerance, impaired cardiac function, a central fat redistribution, increased peripheral arterial resistance, and an unfavorable lipid profile. These effects have been found to be reversed with appropriate replacement therapy with recombinant human growth hormone. We plan to utilize several experimental systems to further investigate the role of growth hormone (GH) in maintaining cardiovascular health. In particular, we would like to further understand the interaction of GH with Plasminogen-activator-inhibitor-1 (a major activator of the fibrinolytic system) as well as the role of GH in the maintenance of vascular function.

ELIGIBILITY:
Inclusion Criteria:

* Adult between the ages of 18 and 65
* Documented Growth Hormone Deficiency as defined by a peak Growth Hormone during a GHRH-Arginine Stimulation test not exceeding 9.5 ng/ml

Exclusion Criteria:

* Personal history of cardiovascular disease (previous myocardial infarction or known coronary artery disease) or diagnosis of heart disease between study visits.
* Personal history of diabetes mellitus or development of diabetes between study visits.
* Initiation of an anti-cholesterol medication or anti-hypertensive between baseline and follow-up study visit.
* Initiation of regular tobacco use between baseline and follow-up study visit.
* Pregnancy or nursing
* Current daily use of any drug known to affect the fibrinolytic system: Aspirin, Aggrenox, Plavix, Persantine, Ticlid, Pletal, Trental, Lovenox, Coumadin, Agrylin, and Hydroxyurea.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26
Dates: Start 2005-08; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doug Vaughan, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Devin JK, Blevins LS Jr, Verity DK, Chen Q, Bloodworth JR Jr, Covington J, Vaughan DE. Markedly impaired fibrinolytic balance contributes to cardiovascular risk in adults with growth hormone deficiency. J Clin Endocrinol Metab. 2007 Sep;92(9):3633-9. doi: 10.1210/jc.2007-0609. Epub 2007 Jun 19. PMID 17579195